CLINICAL TRIAL: NCT05498688
Title: The Acute Effect of a Low-carbohydrate Meal on the Plasma Fatty Acid Composition in Patients With Type 2 Diabetes
Brief Title: The Acute Effect of Low-carb Diet on the Plasma Fatty Acid Composition in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Karina Vejrum Sørensen, Nutrition consultant, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S-20220003
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes
Keywords: Low carbohydrate diet; LCD; Plasma FA composition; Free fatty acids; Cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carbohydrate (Experimental): The intervention meal is a low-carbohydrate meal composed of 15 E% carbohydrates, 20 E% protein and 65 E% fat
  Interventions: Dietary Supplement: Low carbohydrate
- Control meal (No Intervention): The control meal is a regular diabetes meal according to the official Danish dietary guidelines composed of 50 E% carbohydrates, 20 E% protein and 30 E% fat

INTERVENTIONS:
Dietary Supplement: Low carbohydrate — Participants will have a low carbohydrate meal
  Other Names: LCD
  Arms: Low carbohydrate

SUMMARY:
The investigators wishes to investigate the acute effect of a low carbohydrate meal on the plasma fatty acid (FA) composition compared with a control meal in a cross-over study of patients with type 2 diabetes (T2D).

In two trial days 12 participants with T2D will either have a low carbohydrate meal or control meal, measurements will be performed at baseline and continuously over 5 hours.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is the most common metabolic disorder worldwide, and with an increasing prevalence T2D has become a major healthcare burden.

Low carbohydrate diet (LCD) has become increasingly popular as a method of improving glycemic control in patients with type 2 diabetes. However, the higher content of especially saturated fat in LCD has raised concerns about harmful effects.

A previous study has shown increase in non esterified fatty acids after a low carbohydrate meal, but it still needs to be investigated how a low carbohydrate meal affects the plasma FA composition.

The aim of this project is to investigate the hypothesis that a single low carbohydrate meal results in an improved plasma FA composition in patients with T2D and that this, at least in part, corresponds to the changes observed after 6 months LCD.

The study will be conducted as a cross-over trial with 12 participants with T2D. The participants will randomly be assigned to either start with the low carbohydrate meal or a control meal with a 2 weeks washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Duration of established type 2 diabetes for more than six months and less than five years, but duration of type 2 diabetes for up to 10 years if the current treatment consists of ≤ 2 oral antidiabetic drugs without insulin.
2. HbA1c in compliance with type 2 diabetes (above 48 mmol/mol), with or without use of glucose-lowering pharmacotherapy, but without need for adjustment of antidiabetic treatment.
3. Stable antidiabetic treatment three months prior to inclusion.
4. Well treated dyslipidemia (LDL cholesterol < 2.5 mmol/l and total cholesterol < 4.5 mmol/l at inclusion) with or without statins.
5. BMI ≥ 25.
6. Age ≥ 18 years.
7. All participants have to understand oral and written Danish.
8. All participants have to sign an informed consent after oral and written information on experimental design.

Exclusion Criteria:

1. Significant comorbidity, including liver disease.
2. A history of cancer < 5 years or current chemotherapy.
3. Other severe co-morbidity that could interfere with study compliance or safety (e.g. previous gastrointestinal operations, liver disease, history of eating disorder, current alcohol overuse or hypoglycemic unawareness).
4. Current treatment with glucocorticoids (systemic).
5. Continuous treatment with steatosis-inducing drugs.
6. Treatment with antibiotics during the last two months before inclusion.
7. Low-carbohydrate diet prior to inclusion, or other restrictive diet.
8. Weight-loss > 10 kg over the last three months before inclusion.
9. Pregnancy or expected pregnancy within the next 6 months.
10. Elevated blood pressure (180/110) with or without antihypertensives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Plasma fatty acid composition | 5 hours
  Quantified as weight percentage (wt%) of total plasma phospholipid FA

SECONDARY OUTCOMES:
Plasma glucose | 5 hours
Serum insulin | 5 hours
Plasma ketones | 5 hours
Plasma free fatty acid | 5 hours
Total cholesterol | 5 hours
LDL cholesterol | 5 hours
HDL cholesterol | 5 hours
Triglycerides | 5 hours
Other lipoprotein fractions | 5 hours
Glucagon Like Peptide 1 (GLP1) | 5 hours
Glucose-Dependent Insulinotropic Polypeptide (GIP) | 5 hours
Cholecystokinin (CCK) | 5 hours
Peptide YY (PYY) | 5 hours
Ghrelin | 5 hours
Subjective appetite | 5 hours
  Visual analog scale - mm. 0 mm - 100 mm. 0 mm = none and 100 mm = very strong

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Højlund, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No